CLINICAL TRIAL: NCT01298999
Title: Randomized Placebo-Controlled Trial of YF476, a Gastrin Receptor Antagonist, in Barrett's Esophagus
Brief Title: Trial of a Gastrin Receptor Antagonist in Barrett's Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Trio Medicines Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAE9648; YFBE-001 (Other: Trio)
Record Dates: First submitted 2011-02-14; First posted 2011-02-18 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's Esophagus; Esophageal Adenocarcinoma; GERD; Acid Reflux
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus; Gastroesophageal Reflux | interventions — YF 476

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- YF476 (Experimental): YF476 (gastrin-receptor antagonist)
  Interventions: Drug: YF476
- Placebo (Placebo Comparator): Placebo pill (identical in appearance to YF476 pills)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YF476 — 25 mg: one capsule to be taken by mouth once daily for 12 weeks.
  Other Names: Netazepide
  Arms: YF476
Drug: Placebo — Matching placebo: one capsule to be taken by mouth once daily for 12 weeks.
  Other Names: Placebo Tablet
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether treatment with an experimental drug called YF476 in patients with Barrett's esophagus reduces the expression of tissue markers that are associated with an increased risk of developing esophageal cancer.

DETAILED DESCRIPTION:
The association between gastro-esophageal reflux disease (GERD) and cancer of the esophagus is well-established. Barrett's esophagus (BE) is a condition in which the lining of the part of the esophagus changes to look like small intestine, and this change occurs in the setting of GERD. Patients with BE are at increased risk for developing esophageal cancer. It is recommended that all patients with BE take medicines called proton pump inhibitors (PPIs), which greatly reduce the acid produced by the stomach, in the hopes of reducing the risk of esophageal cancer. However, by reducing the acid level in the stomach, levels of a hormone called gastrin are increased. There is laboratory data to suggest that gastrin may have effects that actually promote the development of cancer, including esophageal cancer. The investigators previously showed that BE patients with very high gastrin levels are more likely to have either advanced precancerous changes (also called high grade dysplasia) or cancer of the esophagus. As such, the obvious question is raised: does gastrin promote the development of cancer in BE? YF476 is a new drug that blocks the effects of gastrin. Trials in healthy subjects have demonstrated that the drug is safe and well-tolerated. The investigators therefore propose to conduct a randomized placebo-controlled trial of YF476 in patients with Barrett's esophagus. The primary hypothesis is that treatment with YF476 will reduce the expression of tissue markers that are associated with an increased risk of developing esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years, with histologically confirmed diagnosis of Barrett's Esophagus without dysplasia
* Minimum of 1 cm circumferential Barrett's mucosa on endoscopy or at least 2 cm maximal contiguous extent of Barrett's mucosa
* Proton pump inhibitor use at least once daily for at least twelve months prior to enrolment, and stable dose of PPI for the three months before enrolment
* ECOG performance status ≤ 2 and Karnofsky ≥ 60%
* Normal organ and marrow function
* Use of adequate contraception during the study
* Willingness to comply with all treatment and follow up procedures
* Ability to understand and the willingness to sign a written informed consent document
* Up to date with all age appropriate cancer screening tests, as per American Cancer Society guidelines

Exclusion Criteria:

* Histologically confirmed BE with high grade dysplasia, invasive carcinoma of the esophagus, low grade dysplasia
* Prior endoscopic therapy for BE
* History of esophageal or gastric surgery
* History of atrophic gastritis, pernicious anemia, or Zollinger-Ellison syndrome
* Participation in a trial of an investigational medicinal product within the previous 28 days
* Prolonged QTc interval >450 msec
* History of allergic reactions attributed to compounds of similar chemical composition to YF476
* History of baseline findings of: diabetes mellitus requiring insulin therapy; pancreatitis; hepatitis B, hepatitis C or HIV; malabsorption syndrome or inability to swallow or retain oral medicine; major surgery ≤ 28 days prior to enrollment; ECOG performance status ≥ 2; or another cancer within 3 years except for basal carcinoma of the skin or cervical carcinoma in situ; any clinically significant and uncontrolled major morbidity
* Certain medicines and herbal remedies taken during the 7 days before the start of study drug
* Has evidence of cancer at the time of enrolment, or has surveillance tests planned within 21 weeks after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-06; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian A Abrams, MD, MS, Principal Investigator — Columbia University
Locations (2):
- New York Presbyterian Hospital - Columbia, New York, New York, United States
- National Institute for Health Research, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abrams JA, Del Portillo A, Hills C, Compres G, Friedman RA, Cheng B, Poneros J, Lightdale CJ, De La Rue R, di Pietro M, Fitzgerald RC, Sepulveda A, Wang TC. Randomized Controlled Trial of the Gastrin/CCK2 Receptor Antagonist Netazepide in Patients with Barrett's Esophagus. Cancer Prev Res (Phila). 2021 Jun;14(6):675-682. doi: 10.1158/1940-6207.CAPR-21-0050. Epub 2021 Mar 29. PMID 33782049

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects were screen failures. 24 out of 27 subjects were randomized.
Period: Overall Study
Arm/Group | YF476 | Placebo
Started | 13 | 11
Completed | 10 | 10
Not Completed | 3 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Baseline Endoscopy showed low grade dysplasia or indefinite for dysplasia | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | YF476 | Placebo | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.4 (7.2) | 68.6 (6.6) | 66.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 11 | 10 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, white | 13 | 11 | 24
BMI [Mean (Standard Deviation); unit: kg/m2] | 28.9 (4.7) | 26.7 (3.1) | 27.9 (4.1)
Waist circumference [Mean (Standard Deviation); unit: cm] | 95.7 (17.8) | 98.1 (10.9) | 96.8 (14.8)
Current smoker [Count of Participants; unit: Participants] | 0 | 0 | 0
Proton Pump Inhibitor (PPI) frequency [Count of Participants; unit: Participants]
  Once daily | 8 | 6 | 14
  Twice daily | 5 | 5 | 10
Aspirin Use [Count of Participants; unit: Participants] | 3 | 2 | 5
Barrett's Esophagus length [Mean (Inter-Quartile Range); unit: cm] — Maximal Barrett's esophagus length (Prague M) Population: Arms analyzed separately.
  cm
    YF476: number analyzed (Participants) | 13 | 0 | 13
    YF476 | 3 [2 to 4] |  | 3 [2 to 4]
    Placebo: number analyzed (Participants) | 0 | 11 | 11
    Placebo |  | 6 [4 to 9] | 6 [4 to 9]
Hiatal hernia size [Mean (Inter-Quartile Range); unit: cm] — Population: Arms analyzed separately.
  cm
    YF476: number analyzed (Participants) | 13 | 0 | 13
    YF476 | 2 [2 to 4] |  | 2 [2 to 4]
    Placebo: number analyzed (Participants) | 0 | 11 | 11
    Placebo |  | 4 [3 to 5] | 4 [3 to 5]
Serum gastrin [Mean (Standard Deviation); unit: pmol/L] — At baseline
  pmol/L | 60.3 (41.7) | 51.8 (29.1) | 56.4 (36.0)
Plasma CgA [Mean (Standard Deviation); unit: nmol/L] — At baseline
  nmol/L | 12.9 (17.2) | 9.1 (5.0) | 11.2 (13.0)

OUTCOME MEASURES:

1. Primary Outcome: Mean Ki67 Expression
Description: The study is designed to examine change in tissue Ki67 expression, a marker of cellular proliferation.
Time Frame: Up to 3 months from baseline
Population: Analysis limited to those who completed study (10 subjects in the intervention group and 10 subjects in the placebo group).
Measure: Mean (Standard Deviation); unit: cells/mm2
Arm/Group | YF476 | Placebo
Number analyzed (Participants) | 10 | 10
cells/mm2 | 35.6 (620.7) | 307.8 (640.3)

2. Primary Outcome: Number of Participants That Experienced Change in Any Biomarker Expression
Description: Participants with changes in gene expression were assessed by RNA-sequencing (i.e., sample has sufficient RNA for analysis) between baseline and up to 3 months are tallied.
Time Frame: Up to 3 months from baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | YF476 | Placebo
Number analyzed (Participants) | 10 | 10
Participants | 10 | 9

3. Secondary Outcome: Number of Participants That Experienced Adverse Events
Description: A measure of safety and tolerability. Participants with recorded adverse events were tallied. The events include any adverse events and/or severe adverse events.
Time Frame: Up to 4 months from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | YF476 | Placebo
Number analyzed (Participants) | 13 | 11
Participants
  Serious Adverse Event | 1 | 0
  Any Adverse Event | 10 | 7

ADVERSE EVENTS:
Time Frame: Throughout the course of treatment and up to four weeks after completion of the study drug course or placebo course - an average of 4 months.
Arm/Group | YF476 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/11
Other Adverse Events (participants affected / at risk) | 10/13 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | YF476 (N=13) | Placebo (N=11)
Scrotal abscess (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | YF476 (N=13) | Placebo (N=11)
Diarrhea (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Rectal bleeding (Gastrointestinal disorders) | 1 | 1
Acid reflux (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 3
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Dizziness (Nervous system disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Epistaxis (General disorders) | 0 | 1
Hypoglycemia (Endocrine disorders) | 1 | 0
Mouth ulcer (General disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Relatively small sample size; study enrollment was limited to Barrett's esophagus without dysplasia, limited analysis of treatment related to later stages of disease progression; only one dose was tested which limits possibility that higher doses would have been more bioactive in Barrett's esophagus tissue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT01298999/Prot_SAP_000.pdf